CLINICAL TRIAL: NCT03331653
Title: Effectiveness of Dry Needling and Ischemic Compression in the Sternocleidomastoid, on Cervical Motor Control in Patients With Cervical Pain, Versus Placebo Technique and Ischemic Compression, Randomized Trial.
Brief Title: Effectiveness of Dry Needling and Ischemic Compression in Sternocleidomastoid, on Cervical Motor Control in Patients With Cervical Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Aida Martín Rodríguez, Degree Physiotherapy, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEIM/HU/2017/15
Record Dates: First submitted 2017-11-01; First posted 2017-11-06 (Actual); Last update posted 2018-06-13 (Actual); Status verified 2018-06

CONDITIONS: Cervical Pain
Keywords: Cervical Pain; Motor Control; Sternocleidomastoid; Dry Needling
MeSH Terms: conditions — Neck Pain | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial (RCT) with two groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: Double-blind, masking the patient and the outcomes assesor. A simple randomization will be performed with Epidat software.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Needling and Ischemic Compression at the Trigger Point (Experimental): Dry Needling and Ischemic Compression at the Trigger Point
  Interventions: Other: Dry Needling and Ischemic Compression at the Trigger Point
- Intervention at 1.5 cm from the Trigger Point (Active Comparator): Dry Needling and Ischemic Compression at 1.5 centimeters from the Trigger Point
  Interventions: Other: Dry Needling and Ischemic Compression at 1.5 centimeters from the Trigger Point

INTERVENTIONS:
Other: Dry Needling and Ischemic Compression at the Trigger Point — The intervention consist on dry needling in the active trigger point, and next, do ischemic compression in the same point.
  Arms: Dry Needling and Ischemic Compression at the Trigger Point
Other: Dry Needling and Ischemic Compression at 1.5 centimeters from the Trigger Point — The intervention consist on dry needling at 1.5 centimeters from the active trigger point, and next, do ischemic compression in the same point.
  Arms: Intervention at 1.5 cm from the Trigger Point

SUMMARY:
This study will compare the effect of dry needling on the active trigger point on sternocleidomastoid versus the effect of dry needling at 1.5 centimeters of active trigger point on sternocleidomastoid, both combined with ischemic compression, on cervical pain and cervical motor control short and medium term.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 and 65 years old
* Have pain in the cervical region, which extends from the occipital to the 7th cervical vertebra.
* Have an active trigger point on the sternocleidomastoid.

Exclusion Criteria:

* Present history of trauma in the neck.
* Present cervical radiculopathy
* Present a vestibular pathology
* Previous surgery on the neck or shoulder area
* Having a primary headache diagnosis
* Have received dry needling in the neck in the previous 6 months
* Present cognitive deficit.
* Be pregnant
* Taking anticoagulants.
* Have phobia to the needles (belonephobia).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-11-10 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-06-10 (Actual)

PRIMARY OUTCOMES:
Cervical Pain | Pre-intervention, immediately post-intervention, 1 day, 1 week, 1 month
  Changes in the level of Cervical Pain.
Cervical Motor Control | Pre-intervention, immediately post-intervention, 1 day, 1 week, 1 month
  Change in the Cervical Motor Control

SECONDARY OUTCOMES:
Cervical Range of Movement | Pre-intervention, immediately post-intervention, 1 day, 1 week, 1 month
  Changes in grades of cervical movement
Coordination of superficial and deep cervical flexor muscles | Pre-intervention, immediately post-intervention, 1 day, 1 week, 1 month
  Changes in the coordination of cervical flexor muscles
Cervical Disability | Pre-intervention,1 month
  Changes in perceived cervical disability

CONTACTS AND LOCATIONS:
Overall Officials: Aida M. Rodríguez, Physiotherapy, Principal Investigator — Investigator; Esther S. Olmo, Physiotherapy, Principal Investigator — Investigator
Locations (1):
- University of Alcalá, Alcalá de Henares, Madrid, Spain